CLINICAL TRIAL: NCT04465448
Title: Evaluation of the Reproducibility of the Measurement of the QSM Signal (Quantitative Susceptibility Mapping)
Acronym: ERESI
Status: Terminated | Type: Observational
Why Stopped: MRI issue.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JSY_2020_25
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2022-12

CONDITIONS: White Matter Hyperintensity; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers
  Interventions: Other: MRI
- group case
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Those included will perform an MRI without injection to obtain the QSM then they will exit the machine and reinstall themselves there to perform the second measurement. They will then change the MRI machine to perform a third measurement

SUMMARY:
Many central nervous system pathologies have an inflammatory component, often associated with an accumulation of disability and more severe tissue damage.

In multiple sclerosis, the inflammatory process is in part characterized by the activation of microglia, an entity of the innate inflammatory system, as well as a breakdown of the blood-brain barrier. During inflammation, activated microglia may contain high levels of iron, characterizing its activated state.

DETAILED DESCRIPTION:
Several MRI imaging tools are known to be highly sensitive to tissue iron content and have become the method of choice to study brain iron, including in a pathological context such as multiple sclerosis.

Quantitative magnetic susceptibility mapping (QSM) is an emerging technique to access non-invasively the iron content in brain tissue. For some years this technique has been used in MS to characterize white matter lesions. Changes in the QSM value of the lesions have made it possible to describe lesions surrounded by an iron ring. Susceptibility MRI has also been proposed to highlight lesions according to their chronology.

The study of reproducibility is of particular importance when using QSM in longitudinal studies or in therapeutic trials. A better understanding of intra- and inter-subject variation in QSM measurements may also allow a more accurate estimate of the number of subjects needed to detect changes in studies. In order to be widely applied to various pathologies, it is therefore necessary to evaluate its reproducibility by estimating the intra- and inter-subject variability for future dissemination in clinical and pharmaceutical studies.

In this project, the invstigators propose to study the reproducibility of QSM acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years old
* Consent to participate in the study
* Beneficiary of a social protection scheme
* Healthy volunteers: Consent to be informed if an unexpected anomaly is revealed by the imagery.
* Patients: With MS defined according to McDonald's revised criteria for spatial dissemination and temporal or clinical or radiological temporal dissemination and who should benefit from MRI in the imaging department

Exclusion Criteria:

* Absolute contraindication to 3T MRI
* Realization of an injected MRI (gadolinium) in the previous year
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* For healthy volunteers: History of neurological pathology or neurological pathology in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participation in the study will be offered to patients with MS (the primary indication for which QSM is studied) as well as to healthy volunteers among staff.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
QSM signal difference at two acquisition times in white matter, on an individual scale | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hhopital fondation adolphe de rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No